CLINICAL TRIAL: NCT03416816
Title: A First-in-Human Phase I Trial to Determine the Safety and the Pharmacokinetic Profile of DSP-0337 in Patients With Advanced Solid Tumors
Brief Title: A Study of DSP-0337 in Patients With Advanced Solid Tumors to Determine the Safety and the Pharmacokinetic Profile
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Alternate development strategy
Sponsor: Sumitomo Pharma America, Inc. (Industry)
Collaborators: Syneos Health (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BBI-DSP0337-101
Record Dates: First submitted 2018-01-18; First posted 2018-01-31 (Actual); Last update posted 2023-11-14 (Actual); Status verified 2023-11

CONDITIONS: Neoplasms
Keywords: DSP-0337
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- DSP-0337 (Experimental): In Part 1 - Up to six dose levels will be investigated in dose-escalating cohorts to identify a maximum tolerated dose (MTD). An additional subset of patients will be treated to assess the effect of food intake on the PK of DSP-0337 administration at the MTD level. Once the recommended Phase 2 dose (RP2D) has been established, patients will be treated with the RP2D to explore preliminary antitumor activity and safety profile.
  Interventions: Drug: DSP-0337

INTERVENTIONS:
Drug: DSP-0337 — DSP-0337 will be administered at the following doses in dose-escalation cohorts, maximum tolerated dose (MTD) for food effect, and recommended phase 2 dose (RP2D) for dose-expansion cohort. Dose 1: 200 mg once daily, Dose 2: 200 mg twice daily, Dose 3: 400 mg twice daily, Dose 4: 600 mg twice daily, Dose 5: 800 mg twice daily, Dose 6: 1000 mg twice daily.

SUMMARY:
This is a Phase 1, open label, multi-center study of orally administered DSP-0337 in adult subjects with advance solid tumors that are refractory to standard treatment, or for whom no effective therapy exists.

DETAILED DESCRIPTION:
The study is comprised of two parts: an initial dose escalation phase utilizing a 3 + 3 design to determine maximum tolerated dose followed by a dose expansion cohort in approximately 30 additional subjects. Study participants will initially receive DSP-0337 orally for 28 days (one cycle of treatment). If clinical benefit is seen, treatment can continue until disease progression.

ELIGIBILITY:
Inclusion Criteria

1. Histologically or cytologically confirmed diagnosis of advanced cancer in patients with solid tumors that are refractory to standard treatment, or for whom no effective therapy exists.
2. Patients must have an Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1.
3. Patients must be at least 18 years of age.
4. Organ function must be adequate as follows:

   * Bone Marrow Reserve: absolute neutrophil count ≥ 1.5 x 10^9/L; platelet count ≥ 100 x 10^9/L; hemoglobin ≥ 9.0 g/dL. Must not have required blood transfusion within 1 week of baseline blood count assessment.
   * Hepatic: bilirubin < 1.5 times the upper limit of normal (ULN); alkaline phosphatase (AP), aspartate transaminase (AST), and alanine transaminase (ALT) < 3.0 x ULN (AP, AST, and ALT < 5 x ULN is acceptable if the liver has tumor involvement).
   * Renal: serum creatinine within normal limits; for patients with levels above the institutional normal value, the calculated corrected creatinine clearance must be ≥ 60 mL/min/1.73 m^2 using the Cockcroft-Gault formula corrected for the body surface area.
5. Toxicities incurred as a result of previous anti cancer therapy (radiation therapy [RT], chemotherapy, or surgery) must be resolved to ≤ Grade 1 except for alopecia and anorexia.
6. Patients must provide written informed consent.
7. Female patients are eligible for the study if they meet the following criteria:

   * Are not pregnant or nursing;
   * Of non-childbearing potential defined as women who have had a hysterectomy, bilateral oophorectomy, medically documented ovarian failure, or are documented postmenopausal (follicle stimulating hormone > 40 mIU/mL); OR,

   Of childbearing potential defined as including women < 55 years of age, even those who have experienced 2 years of amenorrhea; all women should also meet both of the following criteria:
   * A negative serum or urine pregnancy test during Screening,
   * Sexually abstinent or correct and consistent use of one of the following methods of birth control in addition to a male partner using a condom from Screening to 3 months after the last dose of study drug:
   * hormone-containing contraceptive intrauterine device with a failure rate of < 1% per year,
   * cervical cap or diaphragm with a spermicidal agent,
   * tubal sterilization, or
   * vasectomy in male partner. Male patients must agree to sexual abstinence or to consistently and correctly use a condom in combination with one of the above methods of birth control from Screening to 3 months after the last dose of study drug.
8. Life expectancy must be ≥ 3 months.

Exclusion Criteria

1. Has received systemic anti-cancer therapy within the 3 weeks prior to starting the trial.
2. Has received radiotherapy within the 28 days prior to first dose or within 12 weeks for patients with glioblastoma, with the exception of palliative radiotherapy to focal lesions for pain or other symptom control.
3. Has received major surgery within the 4 weeks prior to starting the trial.
4. Has significant inter-current illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with the study requirements.
5. Clinically active known brain metastasis unless the brain metastases have been previously treated and are considered stable. Stable brain metastases are defined as no change on computed tomography (CT) scan or magnetic resonance imaging (MRI) for a minimum of 2 months and no change in steroid dose for a minimum of 4 weeks prior to starting the trial.
6. Is pregnant or lactating.
7. Had prior malignancy other than carcinoma in situ of the cervix or non-melanoma skin cancer, unless that prior malignancy was diagnosed and definitively treated at least 3 years previously with no subsequent evidence of recurrence. If the patient has a medical history of a previous tumor that is not included in this criteria and that the Investigator feels is irrelevant for the objectives of the study, it should be evaluated with the Sponsor or Medical Monitor.
8. Has a corrected QT interval (QTc) > 470 ms or has an electrocardiogram (ECG) with a new abnormal finding that is clinically significant.
9. Has a known clinically significant GI disorder(s) including, but not limited to, inflammatory bowel disease or a history of extensive gastric resection and/or small intestinal resection.
10. Has inability to take oral medications and/or has clinical or radiological diagnosis of bowel obstruction.
11. Had prior treatment with napabucasin (BBI-608).
12. Is not able to avoid the concomitant use of proton pump inhibitors (PPIs) or histamine H2-receptors antagonists, which have long-lasting pH-elevating effects, during DSP-0337 dosing, or avoid the use of antacids until at least 2 hours after dosing.
13. Has a known history of human immunodeficiency virus (HIV) infection, active hepatitis B, or untreated hepatitis C; patients who have completed a course of antiviral treatment for hepatitis C are eligible.
14. Has inability to comply with the protocol or study procedures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2018-05-15 (Actual); Primary Completion 2020-06-15 (Actual); Study Completion 2020-06-15 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose by assessing dose-limiting toxicities (DLTs) | 4 weeks
  Dose escalating cohort
Determination of the Recommended Phase 2 Dose (RP2D) by assessing dose-limiting toxicities (DLTs) | 4 weeks
  Dose escalating cohort

SECONDARY OUTCOMES:
Number of Patients with Adverse Events | 12 months
  Tolerability will be evaluated based on the adverse events (AEs) recorded at each contact with the patient, physical examinations, and the results of laboratory tests. Toxicity will be graded according to the Common Terminology Criteria for Adverse Events (CTCAE), version 4.03.
Pharmacokinetics by assessing drug concentration in blood | 4 weeks
  For food effect, dose escalating cohort
Urine excretion of napabucasin after DSP-0337 administration | 24 hours
  Twenty four-hour urine will be collected and excretion of napabucasin will be evaluated.
Objective response rate (ORR) | 6 months
  Defined as the proportion of patients with a documented complete response or partial response (CR + PR) based on RECIST 1.1.
Time to progression (TTP) | 6 months
  Defined as the time from first dose to the earlier date of assessment of progression by RECIST v1.1.
Progression free survival (PFS) | 12 months
  Defined as the time from first dose to the earlier date of assessment of progression or death by any cause in the absence of progression by RECIST v1.1.

OTHER OUTCOMES:
Exploratory pharmacodynamic evaluation, including phosphorylated STAT3 (pSTAT3) expression level in patient-derived tumor tissue, as potential biomarkers | 12 months

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - Indiana University Health Melvin and Bren Simon Cancer Center, Indianapolis, Indiana
  - Karmos Cancer Center, Detroit, Michigan
  - UT Heatlh San Antonio, San Antonio, Texas
  - Utah Cancer Specialist, West Jordan, Utah